CLINICAL TRIAL: NCT06858930
Title: Assessing the Efficacy of a Preoperative Navigation System in Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Collaborators: Nanyang Orthopedic Hospital (Unknown); Weifang Yidu Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24751-0-02
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Anterior cruciate ligament rupture; ACL reconstruction; Surgical Navigation; Robotic Surgery; Bone Tunnel Footprint Localization Accuracy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Robotic Surgery after Preoperative Navigation vs Traditional Arthroscopic Surgery after Preoperative Navigation
Who Masked: Participant
Masking Description: Throughout the clinical study, efforts should be made to keep participants blinded; however, since participants can learn which surgical instruments they used by obtaining a copy of their hospital records upon discharge, the blinding in this clinical study should be maintained as much as possible until the participants automatically unblind themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Surgery after Preoperative Navigation (Experimental): After planning the preoperative bone tunnel using the navigation system from Naton Robotics, robotic surgery will be performed on the day of the operation.
  Interventions: Procedure: ACL footprint localization after preoperative navigation executed by robotic arm
- Traditional Arthroscopic Surgery after Preoperative Navigation (Active Comparator): After planning the preoperative bone tunnel using the navigation system from Naton Robotics, a senior physician will perform traditional arthroscopic surgery on the day of the operation.
  Interventions: Procedure: ACL footprint localization after preoperative navigation executed by rmanual execution

INTERVENTIONS:
Procedure: ACL footprint localization after preoperative navigation executed by robotic arm — Anterior cruciate ligament (ACL) reconstruction is performed using the preoperative navigation of Naton Robotics, followed by random assignment to either robotic surgery or traditional manual surgery. The difference between the two lies in whether the localization of the ACL footprint is performed by a human or by the robotic arm. The surgical technique is standardized as double-bundle reconstruction.
  Arms: Robotic Surgery after Preoperative Navigation
Procedure: ACL footprint localization after preoperative navigation executed by rmanual execution — Anterior cruciate ligament (ACL) reconstruction is performed using the preoperative navigation of Naton Robotics, followed by random assignment to either robotic surgery or traditional manual surgery. The difference between the two lies in whether the localization of the ACL footprint is performed by a human or by the robotic arm. The surgical technique is standardized as double-bundle reconstruction.
  Arms: Traditional Arthroscopic Surgery after Preoperative Navigation

SUMMARY:
The ACL surgery robot features a preoperative navigation system that enhances the precision of bone tunnel placement. As the first dual-bundle reconstruction surgical robot developed in China, it integrates advanced technology to ensure accurate anatomical alignment. This multi-center study aims to evaluate the robot's effectiveness in improving surgical outcomes and reducing complications, demonstrating the potential of domestic innovations in orthopedic surgery. With its high accuracy in locating bone tunnel footprints, this robot represents a significant advancement in ACL reconstruction techniques.

The trial is designed as a randomized controlled trial (RCT) led by a prospective randomized cohort. The study is initiated by Tsinghua University's long-term professor, Yu Jiakuo, and the product has received China's Class III clinical registration certificate.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperatively, the participant or guardian is willing and able to sign the informed consent form;
2. Patients aged 18 to 80 years (inclusive of 18 and 80 years), regardless of gender;
3. Patients who meet the diagnostic criteria for anterior cruciate ligament (ACL) tear and have no contraindications for implantation;
4. Patients with mature skeletons;
5. Good compliance and willingness and ability to participate in follow-up observations as required.

Exclusion Criteria:

* (1) Participants who have previously participated in other clinical studies of drugs, biological agents, or medical devices but did not meet the primary study endpoint within the specified timeframe; (2) Patients with a known allergy to one or more implanted materials; (3) Patients who are physically frail or unable to tolerate surgery due to other systemic diseases; (4) Presence of active infectious lesions in the knee joint or other parts of the body; (5) Obesity with a BMI > 35; (6) Patients with severe diabetes (acute complications of diabetes, preoperative random blood glucose ≥ 16.7 mmol/L with or without altered consciousness, such as diabetic ketoacidosis, suspected diabetic ketoacidosis, hyperglycemic hyperosmolar state, or lactic acidosis; chronic complications of diabetes leading to severe target organ damage requiring urgent treatment, such as acute cardiovascular and cerebrovascular diseases, renal insufficiency, severe vision loss due to retinal disease, intermittent claudication and ischemic symptoms due to peripheral vascular disease, diabetic foot); (7) Women who are pregnant or breastfeeding; (8) Drug users and substance abusers; (9) Patients who are mentally incapacitated or unable to understand the requirements for participating in the study, making cooperation difficult; (10) Those expected to have poor compliance, unwilling or unable to follow postoperative therapy and/or rehabilitation program instructions; (11) Other comorbid conditions that limit participation in the study, hinder compliance with follow-up, or affect the scientific integrity of the study; (12) Other conditions judged by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2029-01-24 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Bone Tunnel Footprint Localization Accuracy | One week post-surgery
  The localization of bone tunnels is evaluated by comparing the deviation of each tunnel's position from its preoperative planned position at one week post-surgery (hereinafter referred to as "bone tunnel deviation value"). At one week post-surgery, each participant undergoes CT three-dimensional imaging of the knee joint on the surgical side, and the bone tunnel positions of the reconstructed ACL on the femur and tibia are measured. The measurement of the femoral tunnel uses the Bernard and Hertel method, measuring the ratio of the center point of the femoral tunnel relative to the Blumensaat line in terms of the horizontal length and height of the lateral femoral condyle. The measurement of the tibial tunnel uses the Stäubli and Rauschning method, measuring the ratio of the center point of the tibial tunnel in relation to the anterior-posterior and medial-lateral dimensions of the tibial plateau. Each research center has designated researchers review the images, and each tunnel cente

SECONDARY OUTCOMES:
Lysholm score | At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months, researchers assess the Lysholm score of the affected knee joint for each participant.The Lysholm knee score, published in 1982 and revised in 1985, has a total score of 100 points. This scale primarily evaluates daily living and athletic function, scoring eight aspects: limping, pain, support, locking, swelling, instability, stair climbing, and squatting. Among these, pain and instability together account for 50 points. The highest score is 100 points, while the lowest is 0 points.
Relative Anterior Translation of the Tibia | At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months, researchers measure the anterior translation distance of the tibia for both the affected and healthy knee joints of the participants. Each side is measured three times, and the average of these three measurements is taken as the final measurement value for the anterior translation distance of the tibia. The relative anterior translation distance is calculated as the affected tibial anterior translation distance minus the healthy tibial anterior translation distance. Measurements are performed using the Kneelaxity arthrometer.
  Kneelaxity arthrometer is a device used to assess knee joint stability by measuring the anterior translation of the tibia relative to the femur, providing objective data on knee laxity and aiding in the evaluation of knee injuries and surgical outcomes.
Knee Flexion and Extension Angle (Range of Motion) | At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months, researchers use a goniometer to measure the flexion and hyperextension angles of the affected knee joint. Each angle is measured three times, and the average of these three measurements is taken as the final measurement value for each angle.
International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) | At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months, researchers assess the IKDC score for the affected knee joint of each participant. Responses to each item are scored using an ordinal scale, where the answer representing the lowest functional level or highest symptom level receives 0 points. For example, the first item relates to performing the highest level of activity without significant pain; if the response is "I cannot perform any of the above activities due to knee pain," it receives 0 points; if the response is "very vigorous activities, such as jumping or rotating in basketball or soccer games," it also receives 0 points. The second item pertains to the frequency of pain over the past four weeks, where "constant pain" receives 0 points and "no episodes" receives 10 points.
  The scoring method for the IKDC subjective knee function evaluation form involves summing the scores of the above items (the 10th item, "What was your knee function b
Tegner Knee Activity Scale | *At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  The researchers assess the Tegner Knee Activity Scale for the affected knee joint of each participant at preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  Tegner Knee Activity Scale is a scoring system used to evaluate knee function and activity level. The scale scores patients based on the intensity of various activities they have been able to perform over a specific period. The score ranges from 0 to 10, where 0 indicates the inability to perform any activities, and 10 indicates the ability to engage in high-intensity sports, such as competitive-level activities. The Tegner score helps clinicians understand the functional status of the patient's knee and its impact on daily life and sports activities.
Visual Analog Scale (VAS) Score | At preoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months.
  The researchers assess the VAS pain score for each participant at preoperative, 1 week postoperative, 6 weeks postoperative, 3 months postoperative, 12 months, and 24 months, and calculate the improvement rate of the VAS score at 1 week, 6 weeks, and 3 months postoperative.
  Visual Analog Scale (VAS) is a subjective scale used to assess pain intensity. The VAS typically consists of a horizontal or vertical line, usually 10 centimeters long, with endpoints labeled "no pain" (0 points) and "worst imaginable pain" (10 points). Patients score their pain intensity by marking a point on this line.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Chang Gung Hospital., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Results of the Excel table for primary and secondary indicators, with personal information of each patient concealed.